CLINICAL TRIAL: NCT04201691
Title: The Effect of Cervical Mobilization on Tonus, Position Sense and Balance in Multiple Sclerosis Patients
Brief Title: Effect of Manuel Therapy on Tonus, Proprioseption and Balance in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tuba Maden (Other)
Responsible Party: Sponsor-Investigator, Tuba Maden, Principal Investigator, clinical research, Hasan Kalyoncu University
Organization: Hasan Kalyoncu University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2019/106
Record Dates: First submitted 2019-12-12; First posted 2019-12-17 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Postural Balance; Multiple Sclerosis; Cervical Region Disorder Nos; Muscle Tonus; Proprioception
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Participants are grouped randomly. First group and second group are applied different rehabilitation programs. Both of group is rest four weeks. Than second group is applied first group's rehabilitation program and first group is applied second group's rehabilitation program.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional group (Experimental): Conventional group is received conventional rehabilitation program.
  Interventions: Other: classic rehabilitation; Other: classic rehabilitation+mobilization
- mobilization group (Experimental): Mobilization group is received cervical mobilization in addition to conventional rehabilitation program.
  Interventions: Other: classic rehabilitation; Other: classic rehabilitation+mobilization

INTERVENTIONS:
Other: classic rehabilitation — The intervention is conventional rehabilitation that included streching, balance and coordination training. The intervention is applied to participants, manually.
  Other Names: conventional rehabilitation
Other: classic rehabilitation+mobilization — Another intervention is manuel therapy that included gliding technics, rotational technics at cervical region. (in addition to classic rehabilitation). The intervention is applied to participants, manually.
  Other Names: experimental rehabilitation

SUMMARY:
This study is investigates the effect of cervical mobilization on tonus, position sense and balance in patient with multiple sclerosis. Half of participants will received classic rehabilitation program, while the other half will received servical mobilization in addition to classic rehabilitation program.

DETAILED DESCRIPTION:
Cervical region is rich in terms of muscle spindle and reseptors. When this region is touched by physiotherapists, muscle spindles is activited. Thus position sense of joint and balance is developed. Besides, cervical region is parasympathetic area have common relaxed effect. Thus this part can be benefit to regulation of tonus.

ELIGIBILITY:
Inclusion Criteria:

* Expanded Disability Status Scale (EDSS) score was between 2-5,
* According to the modified Ashworth Scale, spasticity is between 1 and 3,
* EDSS Cerebellar System Sub-Scale, Functional System Score ˃1,
* medical condition is stable and no medication changes were made in the last month,
* Vertebro-basillar test negative,
* Not have any other neurological disorder and orthopedic problem to prevent participation in this study
* A score of at least 24 from the Mini Mental Test,

Exclusion Criteria:

* presence of psychiatric or severe cognitive dysfunction,
* pregnancy,
* Having a neurological disease other than MS,
* having had an attack in the last 3 months,
* Botulinum toxin application within the last 6 months,
* participating in physiotherapy program in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Change Modified ashworth scale | Change from Modified ashworth scale at one month
  Modified Ashworth Scale measures resistance during passive soft-tissue stretching and is used as a simple measure of spasticity. The minimum value is 1 and the maximum value is 4. Whether higher scores mean a worse outcome.
Change Berg Balance Test | Change from Berg Balance Test at one month
  The scale rates performance from 0 (cannot perform) to 4 (normal performance) on 14 items. The items explore the ability to sit, stand, lean, turn and maintain the upright position on one leg. A cut-off score of 44 was established as a criterion to identify MS subjects with a high risk of fall based on results in the literature. The minumum value is 0, the maximum value is 56. Whether higher scores mean a better outcome.
Change Dynamic Gait Index | Change from Dynamic Gait Index at one month
  The scale measures the mobility function and the dynamic balance. The eight tasks of this scale include walking, walking with head turns, pivoting, walking over objects, walking around objects and going up stairs. The performance is rated on a 4-point scale. A score of 19 or less has been shown to be related to self-reported falls in people with vestibular disorders. The minimum value is 8, the maximum value is 24. Whether higher scores mean a better outcome.
MyotonPRO | 30 days
  The MyotonPRO is a small, noninvasive hand-held apparatus that provides objective measurements of mechanical muscle properties expressed on a continuous scale. After the device probe is positioned on the skin surface above the muscle being measured, and thereby slightly compressing subcutaneous superficial tissue, it exerts a light quick released mechanical impulse. The subsequent dampened oscillation of the muscle is recorded by an accelerometer and numeric values of muscle parameters are calculated, representing the muscle tone, and biomechanical properties.
Change The timed 25-foot walk | Change from The timed 25-foot walk at one month
  The T25-FW is easy to administer, is useful for a range of walking disabilities, and correlates well with other measures of walking ability. The shortening of the time indicate that the patient recovered.
Change Functional Reach Test | Change from Functional Reach Test at one month
  A yardstick was mounted at the height of the patient's acromion. The patient was asked to stretch their arm parallel to the yardstick with fist closed. Then the patient was asked to lean forward as far a possible without taking a step. The new position of the end of the metacarpal bone was marked and the difference to the starting position was calculated. The mean value of three tries was recorded. The Functional Reach Test is a simple measurement of standing balance. Streched distance is the more longer the more better.
Change Sharpened Romberg | Change from Sharpened Romberg at one month
  Participants were asked to remain standing, on a straight line with one leg behind the other leg, leaving the arms sagging and without impairing the balance. Duration stop criteria were defined as the time it took a participant to dislocate the foot, reach the maximal duration of 30 sec, and contact the observer to avoid falling. Higher scores mean a better outcome.
Change Single Leg Stance Test- Right | Change from Single Leg Stance Test- Right at one month
  Duration of standing was measured in participants standing with dangling arms. Maximal duration of test is 30 sec. Higher scores mean a better outcome.
Change Single Leg Stance Test- Left | Change from Single Leg Stance Test- Left at one month
  Duration of standing was measured in participants standing with dangling arms. Maximal duration of test is 30 sec. Higher scores mean a better outcome.
Change Joint of position sense | Change from Joint of position sense at one month
  Position sense was evaluated with Baseline digital goniometer. Extremity of participant is positioned to target angle and hold it there three seconds before returning to starting position. After returning to the starting position, participants attempted to repeat the previously attained angle. The measurements were repeated three times on both extremities (non-dominant and dominant) with a 30-second rest period separating trials. tests are carried out closed eyes for shoulder, ankle, knee. The angular difference is the more smaller the more better.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)